CLINICAL TRIAL: NCT00176059
Title: Immunoglobulin Induction Therapy in Renal Transplant Recipients on Tacrolimus/Azathioprine or Tacrolimus/MMF: Effects on Th1, Th2, B Cell-/Monokine Responses and Immunoregulatory Autoantibody Levels
Brief Title: Immunoregulatory Effects of Immunoglobulin Induction Therapy in Renal Transplant Recipients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Heidelberg University (Other); Astellas Pharma Inc (Industry); Hoffmann-La Roche (Industry); Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTx-Ig-003
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Renal Failure, Chronic; Renal Transplantation
Keywords: immunoglobulins, intravenous; kidney transplantation; acute rejection; chronic rejection; regulatory autoantibodies; Th1; Th2; B Cell; Monokines; Cytokine promoter gene polymorphisms
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Immunoglobulins, Intravenous; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intravenous immunoglobulins (IVIG)
Procedure: kidney transplantation

SUMMARY:
The aim of this randomized prospective study in renal transplant recipients is to investigate immunological short and long-term effects of an IVIG induction therapy.

Furthermore clinical endpoints (patient and graft survival, incidence of acute and chronic rejection, infectious diseases and graft function) up to three years posttransplant will be analyzed.

DETAILED DESCRIPTION:
Intravenous immunoglobulin (IVIG) preparations are known to be effective in the treatment of various autoimmune and inflammatory disorders due to their immunomodulatory and antiinflammatory properties. It has been demonstrated that IVIG is effective in the treatment of acute vascular rejection and steroid resistant cellular rejection. Furthermore, IVIG has been used to inhibit production of lymphocytotoxic antibodies in highly sensitized patients so that successful cadaveric or living renal transplantation could be performed.

The aim of this randomized prospective study in renal transplant recipients is to investigate immunological short and long-term effects of an IVIG induction therapy on Th1, Th2 and B-cell/monocyte responses, expression of adhesion molecules, costimulatory factors and cytokine receptors and on secretion of immunoregulatory autoantibodies (anti-F(ab)-, anti-F(ab')2G-, anti-hinge autoantibodies). These autoantibodies have been shown to significantly affect the risk of chronic rejection and graft loss.

Furthermore, clinical endpoints (patient and gaft survival, incidence of acute and chronic rejection, infectious diseases and graft function) up to 3 years will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* renal transplant recipients of the Giessen renal transplant unit
* cadaveric and living renal transplants
* first and retransplants

Exclusion Criteria:

* Contraindications against blood-taking (anaemia with hemoglobin < 9,5 g/l, hypotension)
* intravenous immunoglobulin therapy in the last half year before study entry
* Hyperimmunoglobulin therapy for severe CMV infection
* Pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-10; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
patient survival | 1 year / 3 years / 5 years posttransplant
graft survival | 1 year / 3 years / 5 years posttransplant
acute rejection | 1 year
chronic allograft nephropathy | 3 years / 5 years posttransplant

SECONDARY OUTCOMES:
graft function | 1 year / 3 years / 5 years
infectious complications | 1 year
immunoglobulin levels | 1 year
regulatory autoantibody levels | 1 year / 3 years / 5 years
Th1 and Th2 responses | 1 year / 3 years
B-cell/monocyte responses | 1 year / 3 years
Expression of adhesion molecules, costimulatory molecules and cytokine receptors | 1 year / 3 years
proteinuria (quantitative assessment) | 1 year / 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Weimer, Prof. Dr., Principal Investigator — Department of Internal Medicine, University of Giessen, Giessen, Germany
Locations (1):
- Department of Internal Medicine, University of Giessen, Giessen, Germany

REFERENCES:
- [Background] Weimer R, Susal C, Yildiz S, Streller S, Pelzl S, Staak A, Renner F, Dietrich H, Daniel V, Feuring E, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. sCD30 and neopterin as risk factors of chronic renal transplant rejection: impact of cyclosporine A, tacrolimus, and mycophenolate mofetil. Transplant Proc. 2005 May;37(4):1776-8. doi: 10.1016/j.transproceed.2005.02.088. PMID 15919463
- [Background] Weimer R, Zipperle S, Daniel V, Carl S, Staehler G, Opelz G. Superior 3-year kidney graft function in patients with impaired pretransplant Th2 responses. Transpl Int. 1998;11 Suppl 1:S350-6. doi: 10.1007/s001470050496. PMID 9665014
- [Background] Weimer R, Zipperle S, Daniel V, Carl S, Staehler G, Opelz G. Pretransplant CD4 helper function and interleukin 10 response predict risk of acute kidney graft rejection. Transplantation. 1996 Dec 15;62(11):1606-14. doi: 10.1097/00007890-199612150-00014. PMID 8970616
- [Background] Susal C, Dohler B, Opelz G. Graft-protective role of high pretransplantation IgA-anti-Fab autoantibodies: confirmatory evidence obtained in more than 4000 kidney transplants. The Collaborative Transplant Study. Transplantation. 2000 Apr 15;69(7):1337-40. doi: 10.1097/00007890-200004150-00021. PMID 10798750
- [Background] Susal C, Dorr C, Groth J, May G, Opelz G. Pretransplant serum IgA concentration and IgA-anti-Fab autoantibody activity as prognostic indicators of kidney graft survival. Transpl Int. 1994;7 Suppl 1:S586-9. doi: 10.1111/j.1432-2277.1994.tb01450.x. PMID 11271315
- [Background] Susal C, Wiesel M, Staehler G, Groth J, May G, Opelz G. Excellent kidney graft survival in patients with high pretransplant serum IgA concentrations and IgA-anti-Fab autoantibody activity. Transplant Proc. 1995 Feb;27(1):1072-4. No abstract available. PMID 7878810
- [Background] Susal C, Guo ZG, Terness P, Opelz G. Role of anti-IgG autoantibodies in kidney transplantation. Immunol Lett. 1990 Nov;26(2):121-5. doi: 10.1016/0165-2478(90)90133-b. PMID 2269482
- [Background] Susal C, Wiesel M, Schonemann C, Groth J, Carl S, Staehler G, May G, Opelz G. Presensitization and HLA match influence the predictive power of pretransplant serum IgA and IgA-anti-Fab autoantibodies in kidney graft recipients. Transplant Proc. 1997 Feb-Mar;29(1-2):1444-6. doi: 10.1016/s0041-1345(96)00551-9. No abstract available. PMID 9123373
- [Background] Susal C, Kropelin M, Groth J, Wiesel M, May G, Carl S, Staehler G, Opelz G. Protective effect of autoantibodies against the hinge region of human IgG in kidney graft recipients. Transplantation. 1996 Nov 27;62(10):1534-6. doi: 10.1097/00007890-199611270-00032. No abstract available. PMID 8958291
- [Background] Susal C, Kropelin M, Wiesel M, Staehler G, Groth J, May G, Opelz G. Pretransplant IgA-anti-hinge and IgA-anti-Fab autoantibody activity is associated with good kidney graft survival. Transplant Proc. 1995 Oct;27(5):2663-5. No abstract available. PMID 7482869
- [Background] Terness PI, Navolan D, Dufter C, Welschof M, Opelz G. Immunosuppressive anti-immunoglobulin autoantibodies: specificity, gene structure and function in health and disease. Cell Mol Biol (Noisy-le-grand). 2002 May;48(3):271-8. PMID 12030431
- [Background] Terness P, Navolan D, Kohl I, Siedler F, Moroder L, Dufter C, Welschof M, Schneider F, Drugarin D, Opelz G. Role of idiotype-independent anti-IgG autoantibodies in human kidney transplantation: natural anti-F(ab')2 antibodies recognize an IgG1 hinge region epitope. Transplant Proc. 1997 Feb-Mar;29(1-2):1412-4. doi: 10.1016/s0041-1345(96)00614-8. No abstract available. PMID 9123359
- [Background] Terness P, Navolan D, Moroder L, Siedler F, Weyher E, Kohl I, Dufter C, Welschof M, Drugarin D, Schneider F, Opelz G. A natural IgA-anti-F(ab')2gamma autoantibody occurring in healthy individuals and kidney graft recipients recognizes an IgG1 hinge region epitope. J Immunol. 1996 Nov 1;157(9):4251-7. PMID 8892664
- [Background] Tyan DB, Li VA, Czer L, Trento A, Jordan SC. Intravenous immunoglobulin suppression of HLA alloantibody in highly sensitized transplant candidates and transplantation with a histoincompatible organ. Transplantation. 1994 Feb 27;57(4):553-62. PMID 8116041
- [Background] Weimer R, Schweighoffer T, Schimpf K, Opelz G. Helper and suppressor T-cell function in HIV-infected hemophilia patients. Blood. 1989 Jul;74(1):298-302. PMID 2568859
- [Background] Weimer R, Daniel V, Zimmermann R, Schimpf K, Opelz G. Autoantibodies against CD4 cells are associated with CD4 helper defects in human immunodeficiency virus-infected patients. Blood. 1991 Jan 1;77(1):133-40. PMID 1824617
- [Result] Staak A, Renner F, Suesal C, Dietrich H, Rainer L, Kamali-Ernst S, Ernst W, Padberg W, Opelz G, Weimer R. Immunoglobulin induction therapy in renal transplant recipients: Effects on immunoglobulin and regulatory antibody levels. Transplant Proc. 2006 Dec;38(10):3483-5. doi: 10.1016/j.transproceed.2006.10.041. PMID 17175311